CLINICAL TRIAL: NCT05757505
Title: The Efficacy and Safety of the Intracranial Stent (Tonbridge) in Endovascular Treatment of Symptomatic Intracranial Atherosclerotic Stenosis: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Trial
Brief Title: The Efficacy and Safety of Intracranial Stent (Tonbridge) in Endovascular Treatment of Symptomatic Intracranial Atherosclerotic Stenosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ton-Bridge Medical Tech. Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZHTQ 202203
Record Dates: First submitted 2023-02-22; First posted 2023-03-07 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-04

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Intracranial Stent (Tonbridge)
  Interventions: Device: Intracranial Stent (Tonbridge)
- control group (Active Comparator): Wingspan Stent System (Stryker Neurovascular)
  Interventions: Device: Wingspan Stent System (Stryker Neurovascular)

INTERVENTIONS:
Device: Intracranial Stent (Tonbridge) — Endovascular treatment with Intracranial Stent (Tonbridge).
  Arms: experimental group
Device: Wingspan Stent System (Stryker Neurovascular) — Endovascular treatment with Wingspan Stent System (Stryker Neurovascular).
  Arms: control group

SUMMARY:
The purpose of this study is to verify the efficacy and safety of the Intracranial Stent (Tonbridge) in endovascular treatment of symptomatic intracranial atherosclerotic stenosis.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled, non-inferiority clinical trial carried out in 13 centers throughout China. 200 subjects with symptomatic intracranial atherosclerotic stenosis will be treated with the Intracranial Stent (Zhuhai Tonbridge Medical Tech. Co., Ltd.) or the Wingspan Stent System (Stryker Neurovascular) for the expansion of vascular stenosis site. The primary objective of this study is to evaluate the effectiveness and safety of the intracranial stent for endovascular treatment of symptomatic intracranial atherosclerotic stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75;
* Subjects with symptomatic intracranial atherosclerotic stenosis who do not respond to antiplatelet therapy or have poor compensation of collateral circulation and hypoperfusion in the offending vessel blood supply;
* The last onset time of TIA is not limited or the last onset of ischemic stroke is more than 2 weeks;
* The lesion is confirmed to be located in intracranial large arteries, including intracranial segment of the internal carotid artery, middle cerebral artery, intracranial segment of vertebral artery and the basilar artery;
* Target vessel diameter≥2.0mm and ≤4.5mm, lesion length ≤33mm;
* Stenosis degree of intracranial arteries≥70% and ≤99% measured by intracranial angiography (WASID method);
* Intracranial artery stenosis which requiring interventional treatment is a single lesion;
* Subjects have at least 1 atherosclerotic plaque risk factor including hypertension, diabetes mellitus, hyperlipidemia, hyperhomocysteinemia, coronary heart disease, obesity, and smoking history;
* mRS≤2 before enrollment;
* Voluntarily participate in this study and sign the informed consent form, can complete examinations and follow-ups in accordance with the requirements of the protocol during the clinical trial.

Exclusion Criteria:

* Intracranial arterial stenosis caused by non-atherosclerotic lesions: such as arterial dissection, moyamoya disease, vasculitis, active arteritis, etc.;
* Preoperative MRI shows only perforator infarction in the target lesion;
* Preoperative CT or MRI indicates the presence of post-infarct hemorrhagic transformation in the target vascular, or a history of subarachnoid, subdural, and epidural hemorrhage within 30 days before procedure, or the presence of untreated chronic subdural hematoma (≥5mm);
* Severe calcification of target vessels; or target vessel tortuosity or other reasons will make experimental device difficult to reach the target lesion position;
* There is more than 70% stenosis in the distal intracranial large vessels or proximal intracranial and extracranial large vessels of the target vessels, and the presence of unidentified responsible lesions;
* Subjects have a major surgery within 30 days before procedure or intend to be hospitalized for other procedure within 6 months after procedure;
* Intracranial tumors or intracranial arteriovenous malformations, or distal and proximal target vessels combined with aneurysms;
* The target lesion has a history of stent implantation;
* It is suspected that there is severe allergy or contraindication to aspirin, clopidogrel, heparin, contrast media, nitinol and other drugs and devices related to endovascular therapy;
* There is an underlying source of cardiac thrombus, such as atrial fibrillation, left ventricular thrombus, myocardial infarction within 30 days;
* Subjects with an INR > 1.5 or the presence of nonmodifiable bleeding factors;
* Medically uncontrolled severe hypertension (systolic blood pressure > 180 mmHg or diastolic blood pressure > 110 mmHg);
* Severe comorbid conditions or unstable conditions, such as severe heart failure, pulmonary failure, or renal failure (serum creatinine >3.0 mg/dL (264μmol/L)), severe liver insufficiency (ALT or AST >3 times normal), and malignancy;
* Life expectancy is less than two years;
* Women who are pregnant or breastfeeding;
* Subjects unable to complete follow-up due to cognitive impairment, mood disorder, or mental illness;
* Subjects who are enrolled in other clinical trials of drugs/devices and have not yet met the primary endpoint;
* Other circumstances which investigators do not consider are appropriate for intracranial stent treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-11 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of any stroke and death within 30 days | 30±7 days post-procedure
  Stroke includes both ischemic and hemorrhagic stroke. Death includes death due to any cause.

SECONDARY OUTCOMES:
Incidence of in-stent restenosis at 6 months, 12 months, and 24 months | 6 months±60 days, 12 months±30 days, and 24 months±30 days post-procedure
  ISR was defined as greater than 50% stenosis within or immediately adjacent (within 5 mm) of the implanted stent and >20% absolute luminal loss. The degree of intracranial artery stenosis will be measured qualitatively in DSA or CTA examination with WASID method.
Incidence of symptomatic in-stent restenosis at 6 months, 12 months, and 24 months | 6 months±60 days, 12 months±30 days, and 24 months±30 days post-procedure
  Symptomatic in-stent restenosis is defined as ischemic stroke or TIA or other ischemic neurological symptoms which are caused by in-stent restenosis.
Device success rate | intra-procedure
  Device success refers to the successful delivery of the stent to the lesion site through the delivery system during procedure, and the stent is deployed well without bending and displacement.
Procedural success rate | intra-procedure
  Procedural success is defined as stenosis degree less than 30% immediately after procedure.
Ratio of mRS 0-2 at 30 days, 6 months, 12 months, and 24 months | 30±7 days, 6 months±60 days, 12 months±30 days, and 24 months±30 days post-procedure
  Subjects will be evaluated at the follow-up visits with mRS. mRS 0-2 indicates a good prognosis.
Mortality at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of ischemic stroke in the target vessel at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of ischemic stroke in non-target vessel at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of any hemorrhagic stroke at 31 days to 6 months, 6 to 12 months, and 12 to 24 months | 31 days to 6 months, 6 to 12 months, and 12 to 24 months post-procedure
Incidence of device deficiency | After use of device to end of study, assess up to 24 months
  Device deficiency is the unreasonable risk that may endanger human health and life safety in the normal use of medical devices during clinical trials, such as labeling errors, quality problems and malfunctions. Possible device deficiency: labeling errors, product quality problems, design defects, broken sterilization packaging, etc.
Incidence of adverse events (AE) at 30 days, 6 months, 12 months, and 24 months | Through 24 months post-procedure
Incidence of serious adverse events (SAE) at 30 days, 6 months, 12 months, and 24 months | Through 24 months post-procedure

CONTACTS AND LOCATIONS:
Overall Officials: Jianmin Liu, Principal Investigator — Changhai Hospital; Shouchun Wang, Principal Investigator — The First Hospital of Jilin University
Locations (13):
- China (13):
  - The First Affiliated Hospital of Henan Science ＆ Technology University, Luoyang, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Baotou City Central Hospital, Baotou, Neimenggu
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Ningbo First Hospital, Ningbo, Zhejiang
  - Changhai Hospital of Shanghai, Shanghai
  - Shanghai Fourth People's Hospital, Shanghai
  - Tongji Hospitai of Tongji University, Shanghai